CLINICAL TRIAL: NCT01147874
Title: Prevalence of Psoriatic Arthritis in Adults With Psoriasis: An Estimate From Dermatology Practice
Acronym: PREPARE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0881A6-4728; B1801032
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Results first posted 2012-06-21 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-04

CONDITIONS: Psoriasis; Psoriatic Arthritis
Keywords: non-therapeutic; interventional
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic | interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- psoriatic arthritis (PsA) questionnaire (No Intervention)
  Interventions: Procedure: lab draws and imaging

INTERVENTIONS:
Procedure: lab draws and imaging — 1 set of lab draws, imaging consists of radiographic imaging or X-ray, ultrasound and MRI

SUMMARY:
This is a phase 4, multicenter, randomized, non-therapeutic interventional trial in subjects with psoriasis looking for the prevalence of psoriatic arthritis. Subjects will be seen and evaluated by a dermatologist at visit 1 and by a rheumatologist at visit 2. A subset of subjects will then go on to visit 3 for imaging procedures (x-ray, MRI, and ultrasound).

ELIGIBILITY:
Inclusion Criteria:

* Subject is >18 years of age at the time of consent.
* Subject has a confirmed diagnosis of plaque psoriasis by clinical judgment.
* Subject is able to read and complete questionnaires.
* Subjects planning to undergo radiographic evaluation, should not have any contraindications to MRI.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1013 (Actual)
Dates: Start 2010-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (45):
- United States (6):
  - Modern Research Assoc. PLLC, Dallas, Texas
  - Rheumatology Practive of Scott Zashin, MD, Dallas, Texas
  - Center for Clinical Studies Ltd LLP, Houston, Texas
  - Rheumatology Associates of Houston, Houston, Texas
  - Center for Clinical Studies LTD LLP, Webster, Texas
  - Dermatology Associates, Seattle, Washington
- Belgium (2):
  - Universitair Ziekenhuis Gent, Ghent, Belgium
  - Algemeen Ziekenhuis St. Jan, Bruges
- Canada (20):
  - Kirk Barber Research, Calgary, Alberta
  - Stratica Medical, Edmonton, Alberta
  - Rheumatology Research Associates, Edmonton, Alberta
  - The Skin Care Centre-Clinical Trials Unit, Vancouver, British Columbia
  - Winnipeg Clinic, Winnipeg, Manitoba
  - Nexus Clinical Research, St. John's, Newfoundland and Labrador
  - Dermatrials Research, Hamilton, Ontario
  - MAC Research Ind., Hamilton, Ontario
  - K-W Musculoskeletal Research Inc., Kitchener, Ontario
  - Lynderm Research Inc, Markham, Ontario
  - The Toronto Western Hospital-Division of Rheumatology, Toronto, Ontario
  - K.Papp Clinical Research Inc., Waterloo, Ontario
  - Windsor Clinical Research, Windsor, Ontario
  - Medical Office, Windsor, Ontario
  - Innovaderm Research Inc, Montreal, Quebec
  - Institut de Rheumatologie de Montreal, Montreal, Quebec
  - GRMO Inc., Québec, Quebec
  - Centre de Recherche Dermatologique du Quebec metropolitain, Québec, Quebec
  - Diex Research Inc., Sherbrooke, Quebec
  - Clinique Medicale Belvedere, Sherbrooke, Quebec
- Denmark (3):
  - Hudlaegerne, Arhus C
  - Bispebjerg University Hospital, Copenhagen NV
  - Gentofte Hospital, Hellerup
- France (3):
  - CHU de l Archet, Nice
  - Hopital Saint Louis, Paris
  - Hôpital Larrey, Toulouse
- Germany (6):
  - Klinik fuer Dermatologie, Allergologie und Venerologie, Berlin
  - Universitaetsklinikum Erlangen Hautklinik im Internistischen Zentrum, Erlangen
  - Klinikum der Johann Wolfgang Goethe Universitaet, Frankfurt am Main
  - Klinik und Poliklinik fuer Dermatologie und, München
  - Praxis Dres. Bredlich, Rosenbach und Thiele, Osnabrück
  - Klinik und Poliklinik fuer Dermatologie, Regensburg
- Hungary (5):
  - Synexus Magyarorszag Kft., Budapest
  - Debreceni Egyetem Orvos-és Egészségtudományi Centrum, Debrecen
  - Borsod Abauj Zemplen Megyei Korhaz es Egyetemi Oktato Korhaz, Szent Ferenc Korhaz Telephely, Miskolc
  - Miskolci Semmelweis Ignac Egeszsegugyi Kozpont es Egyetemi Oktatokorhaz Nonprofit Kft/Borgyogyaszat, Miskolc
  - Borgyogyaszati es Allergologiai, Szolnok

REFERENCES:
- [Derived] Mease PJ, Gladman DD, Papp KA, Khraishi MM, Thaci D, Behrens F, Northington R, Fuiman J, Bananis E, Boggs R, Alvarez D. Prevalence of rheumatologist-diagnosed psoriatic arthritis in patients with psoriasis in European/North American dermatology clinics. J Am Acad Dermatol. 2013 Nov;69(5):729-735. doi: 10.1016/j.jaad.2013.07.023. Epub 2013 Aug 24. PMID 23981683
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881A6-4728&StudyName=Prevalence%20of%20Psoriatic%20Arthritis%20in%20Adults%20with%20Psoriasis%3A%20%20An%20Estimate%20from%20Dermatology%20Practice

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Participants with psoriasis were observed for 8 weeks.
Period: Overall Study
Arm/Group | All Participants
Started | 1013
Completed | 946
Not Completed | 67
Not completed — Adverse Event | 5
Not completed — Investigator's Request | 1
Not completed — Lost to Follow-up | 25
Not completed — Other | 5
Not completed — Protocol Violation | 5
Not completed — Sponsor's Decision | 2
Not completed — Withdrawal by Subject | 24

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 1013
Age Continuous [Mean (Standard Deviation); unit: Years] | 49.90 (13.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 404
  Male | 609

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Psoriatic Arthritis (PsA) Based on Physical Examination, Medical History and Laboratory Results
Description: PsA: inflammatory arthritis associated with psoriasis that can have an indolent and progressive course. Percentage of participants with PsA was calculated by dividing the number of participants who were classified as positive by the rheumatologist and the total number of participants evaluated using medical history, physical examination and laboratory results as the basis for the diagnosis.
Time Frame: Week 0 through Week 8
Population: Full analysis set (FAS) population included all randomized participants with an answer to the question at Visit 1 (dermatology visit) about previous diagnosis of PsA by a rheumatologist and had an assessment of PsA during the study by a rheumatologist based on medical history, physical examination and laboratory results.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 949
Percentage of participants | 30.0 [27.1 to 33.1]

2. Secondary Outcome: Percentage of Participants With Psoriatic Arthritis (PsA) Based on Physical Examination and Medical History
Description: PsA: inflammatory arthritis associated with psoriasis that can have an indolent and progressive course. Percentage of participants with PsA was calculated by dividing the number of participants who were classified as positive by the rheumatologist and the total number of participants evaluated using medical history and physical examination as the basis for the diagnosis.
Time Frame: Week 0 through Week 8
Population: FAS population included all randomized participants with an answer to the question at Visit 1 (dermatology visit) about previous diagnosis of PsA by a rheumatologist and had an assessment of PsA during the study by a rheumatologist based on medical history, physical examination and laboratory results.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 949
Percentage of participants | 29.6 [26.7 to 32.6]

3. Secondary Outcome: Percentage of Participants With Undiagnosed Psoriatic Arthritis (PsA)
Description: PsA: inflammatory arthritis associated with psoriasis that can have an indolent and progressive course. Primary PsA diagnosis made by rheumatologist based on physical examination, medical history and laboratory test results. Secondary PsA diagnosis made by rheumatologist based on physical examination and medical history only. For both, numerator was number of participants with "No" answer to question concerning previous diagnosis of PsA at Visit 1 (dermatology visit) and were subsequently classified as positive by rheumatologist; denominator was total number of participants evaluated for PsA.
Time Frame: Week 0 through Week 8
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 949
Percentage of participants
  Primary PsA diagnosis | 12.3 [10.3 to 14.6]
  Secondary PsA diagnosis | 12.0 [10.0 to 14.2]

ADVERSE EVENTS:
Time Frame: Visit 2 (rheumatology visit), Visit 3 (imaging studies visit)
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/1013
Other Adverse Events (participants affected / at risk) | 7/1013
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=1013)
Procedural dizziness (Injury, poisoning and procedural complications) | 1
Dizziness (Nervous system disorders) | 1
Claustrophobia (Psychiatric disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.